CLINICAL TRIAL: NCT01976845
Title: Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy of Propofol or Midazolam Versus Placebo for Preoperative Medication in Patients Undergoing Elective Orthopedic Surgery
Brief Title: Efficacy of Propofol or Midazolam Compare to Placebo for Preoperative Medication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Ronald Wender, Chairman, Department of anesthesiology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00025204
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Elective Orthopedic Surgery
Keywords: propofol; midazolam; sedative; anxiolytic; amnesic; recall; Memory; Perioperative outcomes
MeSH Terms: interventions — Midazolam; Propofol; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Propofol (Experimental): Propofol 20 mg IV (2 ml)
  Interventions: Drug: Propofol
- Midazolam (Active Comparator): Midazolam 2 mg IV (2 ml)
  Interventions: Drug: Midazolam
- Saline (Placebo Comparator): Saline 2 ml
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Midazolam — Midazolam (20mg) 2 ml IV, in the pre-op area as a premedication
  Other Names: VERSED
  Arms: Midazolam
Drug: Propofol — Propofol (20mg) 2 ml IV, in the pre-op area as a premedication
  Other Names: Diprivan
  Arms: Propofol
Drug: Saline — Saline 2 ml IV, in the pre-op area as a premedication
  Other Names: Saline solution
  Arms: Saline

SUMMARY:
The purpose of this research is:

To evaluate the sedative (reduces irritability or agitation), anxiolytic (reduces anxiety), and amnesic (produces temporary lack of recall) effects of propofol or midazolam when administered for preoperative medication (before administration of drugs that will put patient to sleep) in comparison to placebo. This study is to test whether the use of the pre-anesthesia medication measurably reduces anxiety in comparison to receiving no pre-anesthesia medication prior to orthopedic procedures.

To assess the effect of propofol in comparison to placebo and midazolam on the ability to recall (memory of):

* when the doctor places the mask on patient's face prior to going to sleep
* recall of 2 pictures
* on your satisfaction with the anesthesia as well as postoperative side effects in post-anesthesia care unit (PACU) e.g., nausea ,vomiting and sedation.

DETAILED DESCRIPTION:
The role of anxiolytic premedication in the ambulatory surgical population is frequently debated. Anesthesiologists may consider the administration of anxiety-reducing drugs unnecessary when anxiety levels are low in outpatients presenting for minor surgery. However, the previous study reports that up to 80% of outpatients expressed a preference for a combination of anxiety-reducing and hypnotic premedication before surgery (1-4). In addition to anxiolysis, goals of anxiolytic premedication include sedation, amnesia, improved patient cooperation, and/or improved patient satisfaction. Intravenous (IV) midazolam is the most commonly used premedicant in the ambulatory setting due to its rapid onset, and short half-life (2,3,5), but its residual effects in the immediate postoperative period may contribute to postoperative sedation, as well as to delayed recovery and discharge-readiness after brief outpatient surgery. Furthermore, White et al. (6) noted that the slope of the dose-response curve for sedation was much steeper with midazolam compared with diazepam, which suggests that midazolam may possess a smaller margin of safety and greater need for careful titration to achieve the desired clinical end-point without untoward side effects.

Propofol has become the IV (intravenous) anesthetic of choice for ambulatory anesthesia because of its excellent recovery profile (7). Clinical experience with propofol in the ambulatory setting suggests that its use is associated with less residual sedation and lower incidence of postoperative nausea and vomiting (PONV) (8). However, there are some undesirable side effects associated with propofol including pain on injection, cardiovascular and respiratory depression, and occasional excitement on emergence from anesthesia (9). Practically, small doses of propofol (10-20 mg IV) have been used as an anxiolytic/sedative medication.

To date, there is only one study that has evaluated propofol versus midazolam versus placebo as premedication (10). In this study, the authors stated that propofol (0.4 mg/kg IV) had anxiolytic effects comparable in magnitude and duration to midazolam (0.04 mg/kg IV) with less memory impairment, respiratory depression and dizziness. However, they did not assess the efficacy of propofol and midazolam as a premedication on the recovery profiles and patient's satisfaction in their study. Compared to placebo and propofol, midazolam was associated with more frequent respiratory depression and significant impairment of anterograde explicit memory. Both propofol and midazolam helped relieve anxiety and lowered blood pressure (compared to baseline) but both were associated with greater dizziness scores (P<0.001, compared to placebo).

They concluded that Propofol had an anxiolytic effect comparable in magnitude and duration to that of midazolam with less memory impairment, respiratory depression and dizziness.

Propofol appears to be an economical, effective and safe alternative to midazolam for treating pre-anesthesia anxiety, and especially to be used for induction of anesthesia (10). (This sentence is not clear).

Therefore, we designed this randomized, double-blind, and placebo-controlled study to evaluate propofol as a premedication and to see if it:

* produces comparable anxiolytic effects to midazolam when compared to placebo, but with less memory impairment
* facilitates early recovery profile
* improves patient's satisfaction with the induction and early recovery from anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to sign an informed consent document
* No allergies to midazolam or propofol
* 18 - 70 years of age
* American Society of Anesthesiologists (ASA) Class I-III adults of either sex

Exclusion Criteria:

* Patients with known allergy, hypersensitivity or contraindications to midazolam, propofol, anesthetic or analgesic medications
* Patients with clinically-significant medical conditions, such as brain, heart, kidney, endocrine, or liver diseases
* Pregnant or lactating women
* Subjects with a history of alcohol or drug abuse within the past 3 months
* Patients chronically using sedative, anxiolytic drugs prior to the surgery
* Morbid obesity (BMI >40 kg/m2)
* Patients who are agitated or confused prior to receiving the drug ( verbal rating scale [VRS] greater then 6)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H Wender, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prior to the day of surgery, potential study patients received a packet of materials (initial patient contact letter, a HIPAA information sheet, and the IRB approved informed consent form) from their surgeon. Patients who were interested in participating in the study were asked to bring the materials to the hospital on the day of surgery.
Pre-assignment Details: Randomization assignment was generated with a 1:1:1 allocation ratio using a computer software program.
  The randomization number specifying the study medication was placed in sealed envelope and given to a non-participating anesthesiologist on the day of the scheduled procedure after completing the patient's preoperative assessment.
Period: Overall Study
Arm/Group | Propofol | Midazolam | Saline
Started | 48 | 48 | 43
Completed | 40 | 40 | 40
Not Completed | 8 | 8 | 3
Not completed — Physician Decision | 8 | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol | Midazolam | Saline | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (13) | 51 (15) | 49 (14) | 51 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 17 | 15 | 56
  Male | 16 | 23 | 25 | 64
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 40 | 120
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg^m2] | 28 (5) | 28 (6) | 28 (5) | 28 (5)

OUTCOME MEASURES:

1. Primary Outcome: Scores on the Verbal Rating Scale For Anxiety
Description: Using the verbal rating scale (VRS) for anxiety (0= none to 10 = extremely nervous)
Time Frame: one day
Measure: Mean (Standard Deviation); unit: Scores on a Scale (0-10)
Arm/Group | Propofol | Midazolam | Saline
Number analyzed (Participants) | 40 | 40 | 40
Scores on a Scale (0-10) | 1.8 (1.8) | 2.3 (2.1) | 2.8 (2.1)

2. Secondary Outcome: Scores on the Verbal Rating Scale For Sleepiness (Sedation)
Description: Using the verbal rating scale (VRS) for anxiety (0= none to 10 = extremely sleepiness)
Time Frame: one day
Measure: Mean (Standard Deviation); unit: Scores on a Scale (0-10)
Arm/Group | Propofol | Midazolam | Saline
Number analyzed (Participants) | 40 | 40 | 40
Scores on a Scale (0-10) | 4.6 (2.5) | 5.2 (2.3) | 2.5 (2.4)

3. Secondary Outcome: Produces Amnesia(Memory Recall)
Description: Ability to recall (memory of):
  •recall of 2 pictures
Time Frame: one day
Population: Subjects who recall the picture
Measure: Number; unit: participants
Arm/Group | Propofol | Midazolam | Saline
Number analyzed (Participants) | 40 | 40 | 40
participants | 30 | 12 | 38

ADVERSE EVENTS:
Time Frame: up to 24 hours
Description: The study lasted the day of the anesthesia procedure.
Arm/Group | Propofol | Midazolam | Saline
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No